CLINICAL TRIAL: NCT02483650
Title: The Registry of Hyperbaric Oxygen Therapy Treated Patients
Brief Title: Hyperbaric Oxygen Therapy Registry
Acronym: HBOTR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: U.S. Wound Registry (Other)
Collaborators: Undersea and Hyperbaric Medical Society (UHMS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CDR004
Record Dates: First submitted 2015-05-28; First posted 2015-06-29 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Air or Gas Embolism; Carbon Monoxide Poisoning; Clostridial Myositis and Myonecrosis (Gas Gangrene); Crush Injury, Compartment Syndrome & Other Acute Traumatic Ischemias; Decompression Sickness; Peripheral Arterial Insufficiency and Central Retinal Artery Occlusion; Severe Anemia; Intracranial Abscess; Necrotizing Soft Tissue Infections; Osteomyelitis (Refractory); Delayed Radiation Injury (Soft Tissue and Bony Necrosis); Compromised Grafts and Flaps; Acute Thermal Burn Injury; Idiopathic Sudden Sensorineural Hearing Loss
MeSH Terms: conditions — Embolism, Air; Carbon Monoxide Poisoning; Anthrax; Gas Gangrene; Crush Injuries; Compartment Syndromes; Decompression Sickness; Retinal Artery Occlusion; Anemia; Osteomyelitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the Hyperbaric Oxygen Therapy Registry (HBOTR) is to provide real world patient outcome and side effect information from electronic health records submitted to a specialty specific hyperbaric registry as part of "Stage 2 of Meaningful Use," including data provided to meet PQRS requirements via the registry's QCDR mission.

Goals include understanding the value of HBOT among patients treated for a variety of conditions in relation to the frequency and severity of HBOT side effects. While randomized, controlled trials can establish the efficacy of treatments like HBOT, because they routinely exclude patients with co-morbid conditions common to those patients seen in usual clinical practice, the results of RCTs are usually non-generalizable. Real world data can be used to better understand the effectiveness of HBOT among typical patients, as well as the risks associated with treatment.

DETAILED DESCRIPTION:
The goal of the Hyperbaric Oxygen Therapy Registry (HBOTR) for Wounds is to provide comparative effectiveness data for patients and to understand whether clinical practice guidelines are followed in the use of HBOT.

Hyperbaric Oxygen Therapy (HBOT) is the use of oxygen at greater than one atmosphere (sea level) pressures and is administered by placing the entire patient in a pressurized vessel and having the patient breathe 100% oxygen. The minimum treatment pressure with evidence to support its use among the conditions approved by the Undersea and Hyperbaric Medical society is 2.0 atmospheres absolute (2 ATA) which is an inspired partial pressure of oxygen of approximately 1,520 mmHg. Hyperbaric treatments which provide less than 100% inspired oxygen at the treatment pressure and/or which provide an inspired partial pressure of oxygen less than 760 mmHg are not hyperbaric therapy. Topically applied oxygen is not hyperbaric oxygen therapy. Oxygen is a drug with a well-defined dose response curve as well as acute and chronic drug effects. HBOT also has side effects including oxygen toxicity to many organ systems. The physiological effects of hyperbaric oxygen therapy are well studied. Effectiveness in real world patients is the best current option to understand the role of HBOT in wound healing.

Hospital based outpatient wound centers participating in the US Wound Registry agree to provide data as part of quality initiatives and to meet their Stage 2 Meaningful use criteria. The HBOTR is a subset of the USWR (Chronic Disease Registry) data. All patient data from all participating hyperbaric centers are transmitted to the USWR where data are then used as designated for benchmarking, to satisfy the requirements of PQRS for advanced practitioners, and for data needed by the UHMS to respond to governmental agencies. Data used for effectiveness research are HIPAA de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Hyperbaric Oxygen Therapy for any UHMS Approved indication

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients seen at participating hospital based outpatient wound and hyperbaric centers where HBOT was administered.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Outcome of problem treated with HBOT | 12 Months
  Counts by outcome type

SECONDARY OUTCOMES:
Major Amputation in Wagner Grade 3, 4, or 5 Diabetic Foot Ulcers Treated with HBOT | 12 Months
  Scored in % of major amputations
Preservation of Function with a minor amputation among patients with Wagner Grade 3, 4, or 5 Diabetic Foot Ulcers Treated with HBOT | 12 Months
  Scored in % of minor amputations

OTHER OUTCOMES:
Complications or Side Effects among patients undergoing Treatment with HBOT | 12 months
  Scores in % of: otic barotrauma, other barotrauma, central nervous system oxygen toxicity, confinement anxiety, pneumothorax, sudden respiratory distress, visual acuity changes, low blood sugar, and pulmonary oxygen toxicity.
Appropriate use of HBOT in patients treated for a Diabetic foot ulcer | 12 Months
  Score in % of cases with appropriate use